CLINICAL TRIAL: NCT00431860
Title: Subclinical COronary Atheroscleorosis Updated With Coronary cT Angiography (SCOUT Study)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Other Study IDs: B-0606/034-019
Record Dates: First submitted 2007-02-05; First posted 2007-02-06 (Estimated); Last update posted 2007-05-03 (Estimated); Status verified 2007-05

CONDITIONS: Coronary Atherosclerosis
Keywords: Coronary atherosclerosis, Spiral Computed Tomography
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Coronary computed tomographic angiography

SUMMARY:
The purpose of this study is to validate the usefulness of 64-slice multi-detecter computeted tomography as a screening tool in asymptomatic population.

DETAILED DESCRIPTION:
A large proportion of patients with sudden cardiac death or nonfatal myocardial infarction (MI) had no prior symptom, which emphasizes the importance of early detection and treatment of the underlying subclinical coronary atherosclerosis before they happen. However, there are no powerful screening methods to detect subclinical coronary atherosclerosis until recently. Traditional CAD risk factors, treadmill exercise test, and EBCT are known to have limited power to detect subclinical coronary atherosclerosis and predict future cardiac events.

Coronary CT angiography (CTA) depicting detailed coronary artery anatomy in a noninvasive fashion would seem to be already one of the mainstays of diagnostic procedure in symptomatic population. Instead of the probability of significant stenosis, CTA could provide information about the location, burden and characteristics of atherosclerotic plaque per se, which might give additional insight to stratify the risk of future cardiac events and therapy.

In this study, we will evaluate the prevalence and characteristics of subclinical coronary atherosclerosis on CTA and its impact on the management in asymptomatic population. And then, we will develop standardized protocol for the management of subclinical coronary atherosclerosis, and follow for adverse cardiac events.

In phase I study, we will enroll subjects who had undergone CTA and analyze the characteristics of plaques on CTA. Also, we will evaluate the impact of CTA by comparing the performance of secondary test with those who had not undergone CTA evaluation.

In phase II study, we will recruit subjects who had significant coronary stenosis on CTA. If the patients had significant stenosis, they will undergo coronary angiography to confirm the severity of stenosis. If they had coronary artery stenosis more than 75%, they will receive percutaneous coronary intervention with drug-eluting stent (DES). If they had intermediate lesion, their treatment option will be judged by the results of fractional flow reserve test. If they had coronary lesion less than 50%, they will be treated only by medication.

When the patients are eligible for study, investigators will give information about the study and obtain written consent. The presence of chest pain symptom will be screened with Rose questionnaire. Medical history and physical examination will be performed, and baseline laboratory work-up will be performed.

Following above treatment guidelines, all patients will be followed for adverse cardiac events for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic subjects
* 20-75 years
* subjects who had undergone spiral coronary CT angiography for health check-up

Exclusion Criteria:

* typical or atypical chest pain
* serious comorbid conditions(i.e. malignancy)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2005-12; Study Completion 2011-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Huk-Jae Chang, MD, PhD, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang hospital, Sungnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Choi EK, Choi SI, Rivera JJ, Nasir K, Chang SA, Chun EJ, Kim HK, Choi DJ, Blumenthal RS, Chang HJ. Coronary computed tomography angiography as a screening tool for the detection of occult coronary artery disease in asymptomatic individuals. J Am Coll Cardiol. 2008 Jul 29;52(5):357-65. doi: 10.1016/j.jacc.2008.02.086. PMID 18652943